CLINICAL TRIAL: NCT00994981
Title: Does Pretreated Magnesium Protect Against Reperfusion Injury in Liver Transplanted Patients?
Brief Title: Magnesium Administration in Liver Transplantation and Reperfusion Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong Eun Kim, Department of Anesthesiology, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Mg-study; Mg-study-1
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Living Donor Liver Transplantation; Reperfusion Injury
Keywords: magnesium and reperfusion injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Magnesium; Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- magnesium (Experimental): Using a table of random numbers, the patients were randomized to receive magnesium solution or normal saline. Allocation concealment was ensured using sequentially numbered, sealed opaque envelopes. Immediately after patient's arrival in the operating room, an anesthesiologist who was not involved in this study opened the envelopes and prepared the study solution outside the operating room.
  Interventions: Drug: magnesium
- normal saline (Placebo Comparator): Using a table of random numbers, the patients were randomized to receive magnesium solution or normal saline. Allocation concealment was ensured using sequentially numbered, sealed opaque envelopes. Immediately after patient's arrival in the operating room, an anesthesiologist who was not involved in this study opened the envelopes and prepared the study solution outside the operating room.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: magnesium — Thirty minutes after the beginning of the anhepatic phase, the patients were received a magnesium solution (MgSO4 25 mg•kg-1 mixed in 100 ml of normal saline) over 20 minutes. A resident anesthesiologist, who was blinded to the group assignment, performed intravenous administration of the study solution and assessed study outcomes.
  Other Names: magnesium sulfate
  Arms: magnesium
Drug: normal saline — Thirty minutes after the beginning of the anhepatic phase, the patients were received 100 ml of normal saline over 20 minutes. A resident anesthesiologist, who was blinded to the group assignment, performed intravenous administration of the study solution and assessed study outcomes.
  Other Names: N/S
  Arms: normal saline

SUMMARY:
The purpose of this study is to evaluate the effect of intravenous magnesium infusion before reperfusion with employing some clinical parameters including blood lactate levels, because the intraoperative changes in the blood lactate levels after hepatic allograft reperfusion served as an accurate predictor of the initial graft function in living donor liver transplantation.

DETAILED DESCRIPTION:
Clinically significant hemodynamic deterioration occurs immediately after reperfusion of the grafted liver by unclamping of the portal vein. Profound hypotension, bradycardia, systemic vasodilation, and a decrease in cardiac output have been reported, and this is described as postreperfusion syndrome (PRS). This hemodynamic instability usually requires adequate and aggressive cardiovascular pharmacologic management and fluid support, and recovers slowly over a period of 30 to 60 minutes.Because the severity of PRS correlates with patient and allograft outcome, prevention of its occurrence or attenuation of the hemodynamic changes may improve outcome. However, not much is known about how to protect against this reperfusion injury.

Reperfusion injury also occurs in myocardial infarction, ischemic spinal cord injury and stroke. Recent experiments have shown protective effects of magnesium to reduce the reperfusion injury of these conditions. Magnesium administration may provide cellular protection during ischemia and reperfusion with stabilizing the cellular transmembrane potential, suppressing excessive cellular calcium influx and energy demand.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for elective living donor liver transplantation

Exclusion Criteria:

* pediatric patients
* re-transplantation
* renal dysfunction
* cardiovascular disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
blood lactate level | at 10 minutes after the beginning of the anhepatic phase and at 10, 30, 60 and 120 minutes after reperfusion

SECONDARY OUTCOMES:
aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin and creatinine level | preoperatively and on POD 1 and POD 5

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Choi, professor, Principal Investigator — Department of Anesthesiology and Pain Medicine, School of Medicine, The Catholic University of Korea, Seoul Saint Mary's Hospital
Locations (1):
- The Catholic University of Korea, Seoul Saint Mary's Hospital, Seoul, South Korea